CLINICAL TRIAL: NCT05713955
Title: Evaluation of Effectiveness and Safety of Autologous BioMatrix OBSiDiAN to Enhance a Stapled Circular Esophagogastric Anastomosis After Ivor Lewis Esophagectomy, a Phase II Study.
Brief Title: OBSiDiAN in a Stapled Circular Esophagogastric Anastomosis After Ivor Lewis Esophagectomy
Acronym: Obsidian ph II
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Vivostat (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-09974
Record Dates: First submitted 2021-11-08; First posted 2023-02-06 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Anastomotic Leak Esophagus
Keywords: anastomotic leakage; esophageal cancer surgery; autologous biomatrix
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- study group (Experimental): For the study group, a unit of autologous BioMatrix OBSiDiAN will be produced. Blood sample (120ml) will be taken after randomization at the ending of the abdominal phase of the surgery. The surgeon will create an esophagogastric anastomosis, after ruling out tension or torsion. Around 1-2ml of autologous BioMatrix OBSiDiAN will be applied on the distal/or proximal resection stump before the stapled anastomose will be created. After firing the standard circular device and creation of a functional anastomosis, a further 2.5-3ml OBSiDiAN must be applied circumferentially on the outside on the anastomosis. Once application is completed, a 30 seconds waiting period is required before putting the esophagus back into the surgical field (study specific). A methylene blue leakage test or other leakage test is performed (standard of care). If there is a leak, the anastomosis will be corrected or the completed procedure has to be done again.
  Interventions: Device: Obsidian

INTERVENTIONS:
Device: Obsidian — To create OBSiDiAN BioMatrix, 120 ml of the the patient's blood is added to the processing unit. The Vivostat® processor unit heats, separates, centrifugates to get the plasma. Batroxobin is added. After again processing, the result is an OBSiDian syringe filled with BioMatrix Obsidian®ASG. This will be applied on the anastomosis

SUMMARY:
Oesophagectomy is very invasive surgery. A leakage at the level of the connection between oesophagus and stomach made during surgery causes a lot more problems and can lead to death. Studies show that the leakage rate sometimes goes up to 40 per cent. The chance of dying if you develop a leak after surgery is 15%, while the overall chance of dying during hospitalisation for this procedure is about 4%. We want to investigate whether the use of this new type of 'glue' (Obsidian®) can reduce the number of leaks. We invite you to participate in a clinical trial with the aim of investigating whether Obsidian® is safe and can reduce the number of leaks after oesophageal surgery in patients with oesophageal cancer. We want to apply a new type of 'glue', Obsidian®, at the level of the new connection between oesophagus and stomach.

DETAILED DESCRIPTION:
STUDY PRODUCT Autologous BioMatrix: Obsidian (medical device class III)

STUDY POPULATION Subjects ≥ 18 years and ≤ 75 years of age scheduled for elective Ivor Lewis esophagectomy for esophageal cancer with a circular stapled intrathoracic esophagogastric anastomosis.

SAMPLE SIZE A total of 90 patients will be included in the study. ENROLEMENT PERIOD Based on an annual number of 70-80 esophagectomies in University Hospital Ghent, we predict an enrolment period of 3 years.

STUDY DURATON Considering a 3 years enrolment period and a 1 year follow up we predict a study duration of 4 years.

PRIMAIRY ANALYSIS

• Anastomotic leak within 30 days post operatively. Anastomotic leak type I, II and III is defined according to the Esophagectomy Complications Consensus Group (ECCG).

ELIGIBILITY:
1. Inclusion criteria Preoperatively

   * Subjects ≥ 18 years and ≤ 75 years who are willing to participate and provide written informed consent prior to any study-related procedures.
   * Subjects with esophageal carcinoma (distal until Siewert II) scheduled for elective minimally invasive Ivor Lewis esophagectomy (cT1-4a,N0-3,M0).

   Intra-operatively

   - Intrathoracic circular stapled esophagogastric anastomosis
2. Exclusion criteria preoperatively

   * Female patients who are pregnant or nursing
   * Participation in another study involving investigational drugs or devices.
   * Use of Avastin within 30 days prior to surgery
   * ASA IV (patient with severe systemic disease that is a constant threat to life)
   * Patients with other malignancies
   * Patients with previous esophageal or gastric surgery
   * Known hypersensitivity to batroxobin and tranexamic acid.
   * HB level < 8 g/dL
   * Patients on medicine containing acetylsalicylic acid not able to stop using the medicine for medical reasons minimum 3 days before taking the blood sampling.
   * Patients on clopidogrel not able to stop clopidogrel for medical reasons 7 days before blood sampling
   * Patients on other platelet aggregation inhibitor therapies not able to stop using the platelet aggregation inhibitor therapies for 3 days before taking the blood sample.

Intra-operatively

* Intra-operative findings that may preclude conduct of the study procedures, such as pleural metastasis, tumor invasion in other organs, …
* Anastomosis preformed differently than the standard of care
* Excessive bleeding (>500 ml) prior to anastomosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak | Absence of anastomotic leak within 30 days post operatively
  Anastomotic leak defined according to the ECCG guidelines type I: local defect requiring no change in therapy or treated medicallly or with dietary modifications type II: localized defect requiring interventional but not surgical therapy, for example, interventional radiology drain, stent or bedside opening and packing or incision type III: localized defect requiring surgical therapy

SECONDARY OUTCOMES:
mortality | from surgery until 30 days post operative
  in hospital mortality
sepsis | from surgery until 30 day post operative
  in hospital sepsis
pneumonia | from surgery until 30 day post operative
  in hospital pneumonia
late anastomotic leakage | from surgery until 90 days post operative
  late anastomotic leakage (ECCG type I, II and III)
stricture | from surgery until 1 year post operative
  stricture of the esophagogastric anastomosis
inflammation WBC | from date of randomisation to postoperative day 5
  post operative inflammation (WBC)
inflammation CRP | from date of randomisation to postoperative day 5
  post operative inflammation (CRP)
ICU stay | from surgery until discharge or until the date of death from any cause, whichever came first, assessed up to 3 months
  length of ICU stay
hospital stay | from surgery until discharge or until the date of death from any cause, whichever came first, assessed up to 3 months
  total hospital stay
thoracic drainage volume | from surgery until removal of thoracic drain within the first week postoperative
  Volume of thoracic drain
thoracic drainage duration | from surgery until removal of thoracic drain within the first week postoperative
  duration of thoracic drain
intra-operative checklist | peroperative
  * Hb > 8 g/dL
  * No tension on the anastomosis
  * No torsion on the anastomosis
  * Complete visibility of the anastomosis
  * Dry operation area
  * Application on the gastric stump
  * Application area of 2 cm proximal and distal of the anastomosis
  * Application completely covering the anastomosis
  * Visible white layer of fibrin sealant
  * Dry for 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Piet Pattyn, Principal Investigator — UZ Gent
Locations (1):
- University Hospital Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Plat VD, Bootsma BT, van der Wielen N, van der Peet DL, Daams F. Autologous Activated Fibrin Sealant for the Esophageal Anastomosis: A Feasibility Study. J Surg Res. 2019 Feb;234:49-53. doi: 10.1016/j.jss.2018.08.049. Epub 2018 Sep 27. PMID 30527497